CLINICAL TRIAL: NCT02902341
Title: The CoCoS Interventional Trial: Caloric Control in Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Elisabeth De Waele, MD, PhD, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/045
Record Dates: First submitted 2016-08-23; First posted 2016-09-15 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Metabolism and Nutrition Disorders
Keywords: Nutrition Therapy
MeSH Terms: conditions — Nutrition Disorders | interventions — Nutrition Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Standard protocol nutrition.
  Interventions: Dietary Supplement: Control
- Nutrition Therapy (Experimental): Resting energy expenditure was measured using indirect calorimetry or calculated. A dietician assessed daily caloric intake during the entire hospitalization. Caloric deficits were calculated. According to a predefined flow-chart protocol, nutritional interventions were launched on different time points. Interventions varied from nutritional modifications to oral supplementation, tube feeding, and parenteral nutrition.
  Interventions: Dietary Supplement: Nutrition Therapy

INTERVENTIONS:
Dietary Supplement: Nutrition Therapy — Nutrition based on measured caloric needs.
  Arms: Nutrition Therapy
Dietary Supplement: Control — Standard protocol nutrition based on calculated caloric needs.
  Arms: Control

SUMMARY:
Background: Malnutrition is widespread among cardiac surgery patients and is independently related to an adverse postoperative evolution or outcome. The investigators aimed to assess whether nutrition therapy (NT) could alter caloric deficit, morbidity, and mortality in patients scheduled for non-emergency coronary artery bypass graft (CABG) or aortic valve surgery.

Methods: 351 patients undergoing either elective CABG or aortic valve surgery were studied. Patients receiving NT were enrolled from January 2013 until December 2014. A historical control group consisted of 142 matched patients. Preoperative nutritional status was evaluated. Resting energy expenditure was measured using indirect calorimetry or calculated. Caloric intake and caloric deficits were assessed. The primary endpoint was to evaluate whether NT could limit caloric deficit (Intake to Need Deviation). A secondary endpoint addressed the potential effect of NT on morbidity and mortality. Patients were followed for one year after surgery.

DETAILED DESCRIPTION:
Background: Malnutrition, often presenting as sarcopenic obesity, is widespread among cardiac surgery patients and is independently related to an adverse postoperative evolution or outcome. Nutritional status and energetic needs or deficits in cardiac surgery patients are poorly documented and undernutrition, though readily modifiable, is an often overlooked condition during hospitalization. The investigators aimed to assess whether nutrition therapy (NT) could alter caloric deficit, morbidity, and mortality in patients scheduled for non-emergency coronary artery bypass graft (CABG) or aortic valve surgery.

Methods: 351 patients undergoing either elective CABG or aortic valve surgery were studied. Patients receiving NT were enrolled from January 2013 until December 2014. A historical control group consisted of 142 matched patients who underwent either type of surgery. In all patients, the NRS 2002 and MUST score were used for evaluating the preoperative nutritional status. Resting energy expenditure was measured using indirect calorimetry or calculated. A dietician assessed daily caloric intake during the entire hospitalization. Caloric deficits were calculated. According to a predefined flow-chart protocol, nutritional interventions were launched on different time points. Interventions varied from nutritional modifications to oral supplementation, tube feeding, and parenteral nutrition. The primary endpoint was to evaluate whether NT could limit caloric deficit (Intake to Need Deviation). A secondary endpoint addressed the potential effect of NT on morbidity and mortality. Patients were followed for one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for conventional non-urgent cardiac surgery type coronary artery bypass graft (CABG) or aortic valve surgery

Exclusion Criteria:

* urgent surgery
* aortic arch surgery or other cardiac surgery procedures requiring sternotomy
* off-pump cardiac surgery
* preoperative hemodynamic instability
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with limitation of caloric deficit (Intake to Need Deviation) during hospital stay after cardiac surgery | 3 months (measured at intervals)

SECONDARY OUTCOMES:
Number of participants with overall survival at 1 year or morbidity (acute heart failure, arrythmia, sepsis or pneumonia) during 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth De Waele, MD, PhD, Principal Investigator — UZ Brussel (Vrije Universiteit Brussel)

IPD SHARING:
Plan to Share IPD: Yes
Publication without revealing patient ID's.

REFERENCES:
- [Background] De Waele E, Mattens S, Honore PM, Spapen H, De Greve J, Pen JJ. Nutrition therapy in cachectic cancer patients. The Tight Caloric Control (TiCaCo) pilot trial. Appetite. 2015 Aug;91:298-301. doi: 10.1016/j.appet.2015.04.049. Epub 2015 Apr 22. PMID 25912786
- [Derived] De Waele E, Nguyen D, De Bondt K, La Meir M, Diltoer M, Honore PM, Spapen H, Pen JJ. The CoCoS trial: Caloric Control in Cardiac Surgery patients promotes survival, an interventional trial with retrospective control. Clin Nutr. 2018 Jun;37(3):864-869. doi: 10.1016/j.clnu.2017.03.007. Epub 2017 Mar 18. PMID 28365080